CLINICAL TRIAL: NCT01446172
Title: Longterm Outcome of Inpatient Cognitive and Behavioral Therapies for Panic Disroder and Agoraphobia
Brief Title: Longterm Outcome of Inpatient Cognitive and Behavioral Therapies for Agoraphobia
Status: Completed | Type: Observational
Sponsor: Modum Bad (Other)
Responsible Party: Sponsor
Other Study IDs: Hedley-1
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Agoraphobia
Keywords: Long term outcome
MeSH Terms: conditions — Agoraphobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cognitive, schema focused, guided mastery, exposure

SUMMARY:
While cognitive therapy and exposure therapy are both proven to be effective for panic disorder and/or agoraphobia when outcome is assenssed up to one year after treatment (Gould et al., 1995) the scientific knowledge about long-term course of these disorders is still scanty. Although several long-term outcome studies have been conducted, the quality of these studies has been questioned.

The aim is to conduct a follow-up study of patients with either panic disorder with history of agoraphobia or agoraphobia without history of panic disorder. the patients were treated in a group format at Modum Bad during the years 1989 to 1997. Four subsamples will be included in the study. Subsample 1 (76 patients treated in 1989 and 1990) received combined cognitive and psychodynamic treatment. Subsample 2 and 3 (46 patients treated in 1992 - 1993) were allocated to either cognitive therapy or guided mastery treatment. Subsample 4 (45 patients treated in 1994 - 1996) received cognitive and schema focused therapy.

In the follow-up study the participants will be requested to complete the same self report measures as they completed at intake, discharge and at previous follow-up times. the participants will also be interviewed using the SCID-I and II as they were at the previous assessments.

The present sample is relatively unique in having received pure psychosocial experimental treatments. The very long term efficacy of cognitive therapy relative to behavioural treatmetns for agoraphobia can be evaluated, and the potential moderating effects of personality disorders can be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Meet the DSM-IV kriteria for either panic disorder, panic disorder with agoraphobia or agoraphobia

Exclusion Criteria:

* psychosis
* dementia
* substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with panic disorder with or without agoraphobia and/or agoraphobia without history of panic disorder who have accepted treatment at an inpatient psychiatric hospital
Sampling Method: Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Modum Bad, Vikersund, Norway